CLINICAL TRIAL: NCT05242549
Title: Application of the Transtheoretical Model to Physical Activity and Health-related Quality of Life Among the Frailty of the Community Elderly
Brief Title: The Application of the Transtheoretical Model to the Frailty Elderly in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, PhD, RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FJU-IRB NO：C110071
Record Dates: First submitted 2022-01-23; First posted 2022-02-16 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Frailty
Keywords: frailty; community elderly; Transtheoretical Model; Physical Activity; Health-related Quality of Life; nutritious
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitness and Nutrition Program for Seniors (Experimental): "Fitness and Nutrition Program for Seniors" includes physical activity training, nutrition education- nursing Information, home-based training, and telecare group care (including APP assistance)
  Interventions: Behavioral: Fitness and Nutrition Program for Seniors
- wait-list (No Intervention): Routine care

INTERVENTIONS:
Behavioral: Fitness and Nutrition Program for Seniors — "Fitness and Nutrition Program for Seniors" uses the Trans-Theoretical Model (TTM) as the framework, which includes physical activity training, nutrition education- nursing Information, home-based training, and telecare group care (including APP assistance).
  Physical activity training comprised muscle training, joint strengthening, and upper and lower limb resistance exercises for older adults who were frail. After administering nutrition education- nursing Information, participants were encouraged to set their own goals to improve their diet. Home-based training and telecare group care depends on the stages of TTM behavior change of the elderly.
  Arms: Fitness and Nutrition Program for Seniors

SUMMARY:
As the age structure shows an aging population while facing physical and mental changes among the frailty of the community elderly. Researchers have successively adopted exercise and nutrition strategies for the frail elderly in the community, to improve their physical function, prevent frailty and increase independent functions. There were researches using technology to improve the physical function of the elderly in the community. The transtheoretical model was a comprehensive model of intentional behavior change that incorporates process-oriented variables to explain and predict how and when the elderly change their health behavior including the elderly adoption healthy behavior. Therefore, the investigators use the Trans-Theoretical Model (TTM) to design the "Fitness and Nutrition Program for Seniors" for participants. From improving physical activity and quality of life, then improving the frailty and restoring overall health.

The research will be a quasi-experimental design. It is expected to invite 84 frailty elderly from the Community-Based Care Center (42 in the experimental group and 42 in the control group). The investigators use the Trans-Theoretical Model (TTM) as the framework, which includes physical activity training, nutrition education- nursing Information, home-based training, and telecare group care, develop the "Fitness and Nutrition Program for Seniors" for 6 months. The primary outcome includes cardiovascular health study (CHS) frailty criteria, short physical performance battery (SPPB), grip strength, Timed Up and Go Test (TUG), the international physical activity questionnaire (IPAQ), and SF-12. The secondary outcome includes BMI, upper arm and calf circumference to measure nutritional status, short from falls efficacy scale international (FES-I), the visual analog scale (VAS) to measure pain, and instrumental activities of daily living (IADL). The investigator will follow the outcome before the intervention, the third month after the intervention, and the sixth month after the intervention. The collected data were analyzed with a generalized estimation equation model of SPSS version 22. Make the participants develop a habit of physical activity combined with a nutritious diet. Let the elderly reduce frail state, increase physical activity, improve health-related quality of life and improve health-related results.

DETAILED DESCRIPTION:
The ageing population of the world is an irreversible international situation because of the rapidly increasing number of elderly populations in the 21st century. As the age structure shows an aging population while facing physical and mental changes among the frailty of the community elderly. Helping them prevent disability and promote health has become the focus of current care. Researchers have successively adopted exercise and nutrition strategies for the frail elderly in the community, to improve their physical function, prevent frailty and increase independent functions. The internet was a simple and fast model to care elderly in the community. There were researches using technology to improve the physical function of the elderly in the community. The transtheoretical model was a comprehensive model of intentional behavior change that incorporates process-oriented variables to explain and predict how and when the elderly change their health behavior including the elderly adoption healthy behavior. Therefore, the investigators use the Trans-Theoretical Model (TTM) to design the "Fitness and Nutrition Program for Seniors" for participants, which includes Home-Based physical activity training, nutrition education, and telecare technology. The investigator use the Trans-Theoretical Model (TTM) to analyze the behavior change process of the participants and to explore important factors during the intervention. From improving physical activity and quality of life, then improving the frailty and restoring overall health.

The research will be a quasi-experimental pretest-posttest design. It is expected to invite 84 frailty elderly from Community-Based Care Center in Shilin Districts in Taipei City, Taiwan (42 in the experimental group and 42 in the control group). The investigators use the Trans-Theoretical Model (TTM) as the framework, which includes physical activity training, nutrition education-nursing Information, home-based training, and telecare group care, developing the "Fitness and Nutrition Program for Seniors" for 6 months for community-dwelling frail older adults. The participants create motivation to start execution through physical activity and nutritional knowledge and provide the experimental group with online home-based training from the three different stages of TTM behavior change. During the intervention period, the investigators will follow the adherence, satisfaction, behavior change stage every month. The investigators use motivation to improve the self-efficacy of the participants and achieve the result of behavior change. Finally, support the frail participants to enter the maintenance phase. The primary outcome includes frailty status (cardiovascular health study (CHS) frailty criteria), Physical Activity (short physical performance battery (SPPB), grip strength, Timed Up and Go Test (TUG), the international physical activity questionnaire (IPAQ)), and Health-related Quality of Life (SF-12). The secondary outcome includes kinanthropometric measures (BMI, upper arm, and calf circumference to measure nutritional status), short from falls efficacy scale international (FES-I), the visual analog scale (VAS) to measure pain, and instrumental activities of daily living (IADL). The investigators will follow the outcome before the intervention, the third month after the intervention, and the sixth month after the intervention. The collected data were analyzed with a generalized estimation equation model of SPSS version 22. The research hopes to promote the health of the frailty participants through FANS in the community. Make the participants develop a habit of physical activity combined with a nutritious diet. Let the participants reduce frail state, increase physical activity, improve health-related quality of life and improve health-related results, and have a healthy life.

ELIGIBILITY:
Inclusion Criteria:

1. ≥65 years old
2. classified as prefrail or frail stage by the Cardiovascular health study (CHS) frailty criteria.
3. Conscious clear and can comply with study procedures.
4. Have a device that enables online communication, and having the ability to operate this device. (Experimental group)

Exclusion Criteria:

1. Diagnosed as unsuitable for physical activity with high risk of acute and chronic diseases, such as neurological impairment, severe cardiovascular or pulmonary disease, persistent joint pain, or severe musculoskeletal impairment or severe musculoskeletal injury, joint or lower extremity surgery within 6 months.
2. severe visual impairment
3. institutionalization
4. Participated in physical activity or nutrition interventional six months ago

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Basic Demographic Health Assessment Form | baseline, pre-intervention(T0)
  Number, age, gender, education level, marriage, living conditions, tobacco and alcohol use, economic status, chronic illness history
Cardiovascular health study (CHS) frailty criteria | baseline, pre-intervention(T0)
  Frailty criteria comprising weak grip of <26.0 kg in men or <18.0 kg in women; walking slower than 0.8 m/s; self-reported exhaustion on more than 3 days/week; unintentional weight loss of >5.0 kg or 10% during the past year; and physical activity <3.75 MET/h in men or <2.5 MET/h in women (lowest quintile of sex-specific baseline values). People fulfilling three or more criteria were classed as frail, those who met one or two as prefrail, and those with no such deficits as robust.
Cardiovascular health study (CHS) frailty criteria | three months after intervention(T1)
  Frailty criteria comprising weak grip of <26.0 kg in men or <18.0 kg in women; walking slower than 0.8 m/s; self-reported exhaustion on more than 3 days/week; unintentional weight loss of >5.0 kg or 10% during the past year; and physical activity <3.75 MET/h in men or <2.5 MET/h in women (lowest quintile of sex-specific baseline values). People fulfilling three or more criteria were classed as frail, those who met one or two as prefrail, and those with no such deficits as robust.
Cardiovascular health study (CHS) frailty criteria | six months after intervention(T2)
  Frailty criteria comprising weak grip of <26.0 kg in men or <18.0 kg in women; walking slower than 0.8 m/s; self-reported exhaustion on more than 3 days/week; unintentional weight loss of >5.0 kg or 10% during the past year; and physical activity <3.75 MET/h in men or <2.5 MET/h in women (lowest quintile of sex-specific baseline values). People fulfilling three or more criteria were classed as frail, those who met one or two as prefrail, and those with no such deficits as robust.
Physical Activity-Short Physical Performance Battery (SPPB) | baseline, pre-intervention(T0)
  SPPB consists of three domains: a Timed 4 m Walk, Balance, and a Chair Sit-to-Stand Test. Each performance measurement was assigned a score from 0 (inability to complete) to 4 (best performance possible). The total of the scores was used to obtain an overall measurement of physical performance. The maximum total score, including all three domains, is 12, and a higher score indicates better physical function.
Physical Activity-Short Physical Performance Battery (SPPB) | three months after intervention(T1)
  SPPB consists of three domains: a Timed 4 m Walk, Balance, and a Chair Sit-to-Stand Test. Each performance measurement was assigned a score from 0 (inability to complete) to 4 (best performance possible). The total of the scores was used to obtain an overall measurement of physical performance. The maximum total score, including all three domains, is 12, and a higher score indicates better physical function.
Physical Activity-Short Physical Performance Battery (SPPB) | six months after intervention(T2)
  SPPB consists of three domains: a Timed 4 m Walk, Balance, and a Chair Sit-to-Stand Test. Each performance measurement was assigned a score from 0 (inability to complete) to 4 (best performance possible). The total of the scores was used to obtain an overall measurement of physical performance. The maximum total score, including all three domains, is 12, and a higher score indicates better physical function.
Physical Activity-Grip Strength | baseline, pre-intervention(T0)
  Grip strength was measured using a dynamometer based on two rounds of measurements for each hand.
Physical Activity-Grip Strength | three months after intervention(T1)
  Grip strength was measured using a dynamometer based on two rounds of measurements for each hand.
Physical Activity-Grip Strength | six months after intervention(T2)
  Grip strength was measured using a dynamometer based on two rounds of measurements for each hand.
Physical Activity-Timed Up and Go Test (TUG) | baseline, pre-intervention(T0)
  Administration of the TUG requires subjects to stand up from a chair, walk 2.44m, turn around, walk back to the chair, and sit down.
Physical Activity-Timed Up and Go Test (TUG) | three month after intervention(T1)
  Administration of the TUG requires subjects to stand up from a chair, walk 2.44m, turn around, walk back to the chair, and sit down.
Physical Activity-Timed Up and Go Test (TUG) | six month after intervention(T2)
  Administration of the TUG requires subjects to stand up from a chair, walk 2.44m, turn around, walk back to the chair, and sit down.
Health-related Quality of Life | baseline, pre-intervention(T0)
  HRQOL was assessed using the Medical Outcomes Survey Short Form-12 questionnaire (SF-12), which consists of eight items representing the following health profile dimensions: general health perception, physical functioning, role functioning-physical, bodily pain, vitality, social functioning, mental health, and role functioning-emotional. Responses are provided using a five- or six-point Likert scale, standardized according to the scoring system. Separate scores are provided for the physical and mental components of health.
Health-related Quality of Life | three months after intervention(T1)
  HRQOL was assessed using the Medical Outcomes Survey Short Form-12 questionnaire (SF-12), which consists of eight items representing the following health profile dimensions: general health perception, physical functioning, role functioning-physical, bodily pain, vitality, social functioning, mental health, and role functioning-emotional. Responses are provided using a five- or six-point Likert scale, standardized according to the scoring system. Separate scores are provided for the physical and mental components of health.
Health-related Quality of Life | six months after intervention(T2)
  HRQOL was assessed using the Medical Outcomes Survey Short Form-12 questionnaire (SF-12), which consists of eight items representing the following health profile dimensions: general health perception, physical functioning, role functioning-physical, bodily pain, vitality, social functioning, mental health, and role functioning-emotional. Responses are provided using a five- or six-point Likert scale, standardized according to the scoring system. Separate scores are provided for the physical and mental components of health.

SECONDARY OUTCOMES:
kinanthropometric measures-BMI | baseline, pre-intervention(T0)
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. We use weight and height will be combined to report BMI in kg/m2.
kinanthropometric measures-BMI | three months after intervention(T1)
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. We use weight and height will be combined to report BMI in kg/m2.
kinanthropometric measures-BMI | six months after intervention(T2)
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. We use weight and height will be combined to report BMI in kg/m2.
kinanthropometric measures-upper arm and calf circumference | baseline, pre-intervention(T0)
  Upper arm and calf circumference were measured to the nearest 0.1 cm using a flexible but nonstretch measuring tape. Upper arm and calf circumference to measure nutritional status
kinanthropometric measures-upper arm and calf circumference | three months after intervention(T1)
  Upper arm and calf circumference were measured to the nearest 0.1 cm using a flexible but nonstretch measuring tape. Upper arm and calf circumference to measure nutritional status
kinanthropometric measures-upper arm and calf circumference | six months after intervention(T2)
  Upper arm and calf circumference were measured to the nearest 0.1 cm using a flexible but nonstretch measuring tape. Upper arm and calf circumference to measure nutritional status
short from falls efficacy scale international (FES-I) | baseline, pre-intervention(T0)
  The 7 items of the FES-I were rated on a 4-point Likert scale with the following possible answers (scores in parentheses): ''not at all'' (1); ''somewhat'' (2); 'fairly' (3); and 'very concerned' (4). If subjects were unable to perform the activity, they were encouraged to respond hypothetically. The range of possible total scores was from 7 to 28, with a high score indicating greater fear of falling.
short from falls efficacy scale international (FES-I) | three months after intervention(T1)
  The 7 items of the FES-I were rated on a 4-point Likert scale with the following possible answers (scores in parentheses): ''not at all'' (1); ''somewhat'' (2); 'fairly' (3); and 'very concerned' (4). If subjects were unable to perform the activity, they were encouraged to respond hypothetically. The range of possible total scores was from 7 to 28, with a high score indicating greater fear of falling.
short from falls efficacy scale international (FES-I) | six months after intervention(T2)
  The 7 items of the FES-I were rated on a 4-point Likert scale with the following possible answers (scores in parentheses): ''not at all'' (1); ''somewhat'' (2); 'fairly' (3); and 'very concerned' (4). If subjects were unable to perform the activity, they were encouraged to respond hypothetically. The range of possible total scores was from 7 to 28, with a high score indicating greater fear of falling.
the visual analog scale (VAS) to measure pain | baseline, pre-intervention(T0)
  ranging from "no pain= 0mm" to "unwilling pain= 100mm". Scores were calculated to the nearest millimetre with a ruler.
the visual analog scale (VAS) to measure pain | three months after intervention(T1)
  ranging from "no pain= 0mm" to "unwilling pain= 100mm". Scores were calculated to the nearest millimetre with a ruler.
the visual analog scale (VAS) to measure pain | six months after intervention(T2)
  ranging from "no pain= 0mm" to "unwilling pain= 100mm". Scores were calculated to the nearest millimetre with a ruler.
Instrumental activities of daily living (IADL) | baseline, pre-intervention(T0)
  IADL is a 15-item questionnaire that assesses recent participation in functional activity. For each item, participants are required to indicate the extent which four statements reflect their recent participation in an activity. Although responses regarding the four statements varied between items, scores generally ranged from 0 ("never") to 3 ("most days" or "at least once weekly"). Total scores, calculated by summing the item scores, range from 0 to 45.
Instrumental activities of daily living (IADL) | three months after intervention(T1)
  IADL is a 15-item questionnaire that assesses recent participation in functional activity. For each item, participants are required to indicate the extent which four statements reflect their recent participation in an activity. Although responses regarding the four statements varied between items, scores generally ranged from 0 ("never") to 3 ("most days" or "at least once weekly"). Total scores, calculated by summing the item scores, range from 0 to 45.
Instrumental activities of daily living (IADL) | six months after intervention(T2)
  IADL is a 15-item questionnaire that assesses recent participation in functional activity. For each item, participants are required to indicate the extent which four statements reflect their recent participation in an activity. Although responses regarding the four statements varied between items, scores generally ranged from 0 ("never") to 3 ("most days" or "at least once weekly"). Total scores, calculated by summing the item scores, range from 0 to 45.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Zhiwuyuan and Fujia Community-Based Care Center, Taipei, Shilin Districts, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barton AC, Sheen J, Byrne LK. Immediate Attention Enhancement and Restoration From Interactive and Immersive Technologies: A Scoping Review. Front Psychol. 2020 Aug 19;11:2050. doi: 10.3389/fpsyg.2020.02050. eCollection 2020. PMID 32973620
- [Background] Gerotziafas GT, Catalano M, Theodorou Y, Dreden PV, Marechal V, Spyropoulos AC, Carter C, Jabeen N, Harenberg J, Elalamy I, Falanga A, Fareed J, Agathaggelou P, Antic D, Antignani PL, Bosch MM, Brenner B, Chekhonin V, Colgan MP, Dimopoulos MA, Douketis J, Elnazar EA, Farkas K, Fazeli B, Fowkes G, Gu Y, Gligorov J, Ligocki MA, Indran T, Kannan M, Kantarcioglu B, Kasse AA, Konstantinidis K, Leivano F, Lewis J, Makatsariya A, Mbaye PM, Mahe I, Panovska-Stavridis I, Olinic DM, Papageorgiou C, Pecsvarady Z, Pillon S, Ramacciotti E, Abdel-Razeq H, Sabbah M, Sassi M, Schernthaner G, Siddiqui F, Shiomura J, Slama-Schwok A, Wautrecht JC, Tafur A, Taher A, Klein-Wegel P, Zhai Z, Zoubida TM; Scientific Reviewer Committee. The COVID-19 Pandemic and the Need for an Integrated and Equitable Approach: An International Expert Consensus Paper. Thromb Haemost. 2021 Aug;121(8):992-1007. doi: 10.1055/a-1535-8807. Epub 2021 Jul 20. PMID 34169495
- [Background] Haider S, Grabovac I, Dorner TE. Effects of physical activity interventions in frail and prefrail community-dwelling people on frailty status, muscle strength, physical performance and muscle mass-a narrative review. Wien Klin Wochenschr. 2019 Jun;131(11-12):244-254. doi: 10.1007/s00508-019-1484-7. Epub 2019 Apr 2. PMID 30941525
- [Background] Jadczak AD, Makwana N, Luscombe-Marsh N, Visvanathan R, Schultz TJ. Effectiveness of exercise interventions on physical function in community-dwelling frail older people: an umbrella review of systematic reviews. JBI Database System Rev Implement Rep. 2018 Mar;16(3):752-775. doi: 10.11124/JBISRIR-2017-003551. PMID 29521871
- [Background] Dent E, Lien C, Lim WS, Wong WC, Wong CH, Ng TP, Woo J, Dong B, de la Vega S, Hua Poi PJ, Kamaruzzaman SBB, Won C, Chen LK, Rockwood K, Arai H, Rodriguez-Manas L, Cao L, Cesari M, Chan P, Leung E, Landi F, Fried LP, Morley JE, Vellas B, Flicker L. The Asia-Pacific Clinical Practice Guidelines for the Management of Frailty. J Am Med Dir Assoc. 2017 Jul 1;18(7):564-575. doi: 10.1016/j.jamda.2017.04.018. PMID 28648901
- [Background] Marston HR, Shore L, White PJ. How does a (Smart) Age-Friendly Ecosystem Look in a Post-Pandemic Society? Int J Environ Res Public Health. 2020 Nov 9;17(21):8276. doi: 10.3390/ijerph17218276. PMID 33182413
- [Background] Nagai K, Miyamato T, Okamae A, Tamaki A, Fujioka H, Wada Y, Uchiyama Y, Shinmura K, Domen K. Physical activity combined with resistance training reduces symptoms of frailty in older adults: A randomized controlled trial. Arch Gerontol Geriatr. 2018 May-Jun;76:41-47. doi: 10.1016/j.archger.2018.02.005. Epub 2018 Feb 13. PMID 29455058
- [Background] Kidd T, Mold F, Jones C, Ream E, Grosvenor W, Sund-Levander M, Tingstrom P, Carey N. What are the most effective interventions to improve physical performance in pre-frail and frail adults? A systematic review of randomised control trials. BMC Geriatr. 2019 Jul 11;19(1):184. doi: 10.1186/s12877-019-1196-x. PMID 31291884
- [Background] Wang L, Chen H, Lu H, Wang Y, Liu C, Dong X, Chen J, Liu N, Yu F, Wan Q, Shang S. The effect of transtheoretical model-lead intervention for knee osteoarthritis in older adults: a cluster randomized trial. Arthritis Res Ther. 2020 Jun 8;22(1):134. doi: 10.1186/s13075-020-02222-y. PMID 32513273
- [Background] Zazzara MB, Vetrano DL, Carfi A, Onder G. Frailty and chronic disease. Panminerva Med. 2019 Dec;61(4):486-492. doi: 10.23736/S0031-0808.19.03731-5. Epub 2019 Jul 30. PMID 31362483
- [Background] Zhang Y, Zhang Y, Du S, Wang Q, Xia H, Sun R. Exercise interventions for improving physical function, daily living activities and quality of life in community-dwelling frail older adults: A systematic review and meta-analysis of randomized controlled trials. Geriatr Nurs. 2020 May-Jun;41(3):261-273. doi: 10.1016/j.gerinurse.2019.10.006. Epub 2019 Nov 6. PMID 31706592
- [Derived] Li PS, Hsieh CJ, Miao NF, Tsai CH, Liu CY, Lin HR, Wu SV, Koh J. Application of the Fitness and Nutrition Program for Seniors (FANS) to improve Physical Activity and Kinanthropometric Measures among Community-Dwelling Older Adults living with Frailty: a Quasi-experimental Study. BMC Geriatr. 2025 Jul 22;25(1):543. doi: 10.1186/s12877-025-06171-6. PMID 40696284
- [Derived] Li PS, Hsieh CJ, Miao NF, Tsai CH, Liu CY, Lin HR, Wu SV, Koh J. Enhancing Frailty Status and Health-Related Quality of Life in Community-Dwelling Frail Older Adults. Gerontology. 2025;71(4):273-291. doi: 10.1159/000543909. Epub 2025 Feb 5. PMID 40552877
- See also: Reablement and older people, Final report of the International Federation on Aging Copenhagen Summit — http://www.ifa-copenhagen-summit.com/wp-content/uploads/2016/04/Copenhagen-Summit-Final-Report.pdf